CLINICAL TRIAL: NCT06068751
Title: The Effectiveness of Aerobic Exercise and Neck Exercises in Pediatric Migraine Treatment: A Randomized Controlled Single-Blind Study
Brief Title: Aerobic Exercise and Neck Exercises in Pediatric Migraine Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Rabia Likos Akpınar, MD in ER, Principal Investigator, Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 139
Record Dates: First submitted 2023-09-22; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Migraine in Children
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise (Active Comparator): Aerobic Exercise
  Interventions: Other: Aerobic Exercise
- Neck Exercises (Active Comparator): Neck Exercises
  Interventions: Other: Neck Exercises

INTERVENTIONS:
Other: Aerobic Exercise — The initial group will receive instructions to increase their moderate to high-intensity physical activity frequency to at least 60 minutes per day (in episodes exceeding 10 minutes) by 50%, with a minimum of three days per week. They will be encouraged to engage in enjoyable and age-appropriate activities, including jogging, brisk walking, swimming, dancing, cycling, as well as sports like basketball, football, and tennis.
  Arms: Aerobic Exercise
Other: Neck Exercises — The second group, focused on neck exercises, will receive guidance from an experienced physiotherapist and their families. The physiotherapist will demonstrate a series of stretching and isometric strengthening exercises for specific muscle groups: upper trapezius, levator scapula, sternocleidomastoid, cervical flexors, and extensors, which have been associated with migraines in prior studies. Each patient will perform 3 sets of 10-15 repetitions for both stretching and isometric strengthening exercises per muscle group, with a 1-minute break between sets. Patients will be advised to maintain a gentle stretch during stretching exercises, avoiding excessive force to prevent discomfort. Static stretching and isometric strengthening exercises will involve holding each position for 5-10 seconds. In the initial week, a reduced set of 5 repetitions will be allowed for adaptation. Throughout the intervention, participants will follow this exercise regimen for 3 days weekly.
  Arms: Neck Exercises

SUMMARY:
This randomized controlled single-blind trial will include 60 pediatric migraine patients. Participants will be divided into two groups: one performing aerobic exercise, and the other conducting neck exercises. Assessments include attack frequency, severity, duration, and neck pain over three months.

ELIGIBILITY:
Inclusion Criteria:

- Pediatric Migraneurs, as per International Classification of Headache Disorders-3 guidelines

Exclusion Criteria:

* individuals with any other concomitant headaches
* those showing findings beyond nonspecific hyperintense areas on cranial Magnetic Resonance Imaging
* patients with systemic diseases other than migraine, such as fibromyalgia
* individuals who had experienced treatment changes or required treatment changes within the last month
* limited mental capacity or psychological illnesses that could hinder their participation in surveys and exercises
* a history of increased attack frequency or severity with previous physical activity program involvement, or a history of trauma to the neck or face
* individuals with a history of a herniated disc in the cervical region or symptoms of cervical radiculopathy

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Migraine Attack Frequency | Baseline, first and third month follow-ups
  The frequency of migraine attacks in patients will be evaluated in days/month.
Migraine Attack Duration | Baseline, first and third month follow-ups
  The duration of attacks in patients will be recorded in hours.
Migraine Attack Severity | Baseline, first and third month follow-ups
  The severity of migraine attacks will be assessed using a visual analog scale, and a score between 0 and 10 will be assigned. A high score indicates more severe attack.
Neck Pain Severity | Baseline, first and third month follow-ups
  The severity of neck pain will be assessed using a visual analog scale, and a score between 0 and 10 will be assigned. A high score indicates severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Orhan Coskun, MD, Study Director — Gaziosmanpaşa Research and Training Hospital
Locations (1):
- Gaziosmanpaşa Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR